CLINICAL TRIAL: NCT00775827
Title: A Randomised, Two-Treatment, Two-Period, Two-Sequence, Single-Dose, Crossover Bioavailability Study on Fenofibrate Formulations Comparing Fenofibrate 160 mg Tablets of Ranbaxy Laboratories With Tricor 160 mg Tablets of in Healthy, Adult, Human Subjects Under Fasting Conditions
Brief Title: Bioequivalency Study of Fenofibrate 160mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 028/FENOF-160/02
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: bioequivalence fenofibrate tablets
MeSH Terms: interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): fenofibrate 160 mg tablets of Ranbaxy Laboratories
  Interventions: Drug: fenofibrate 160 mg tablets
- 2 (Active Comparator): Tricor 160 mg tablets
  Interventions: Drug: fenofibrate 160 mg tablets

INTERVENTIONS:
Drug: fenofibrate 160 mg tablets

SUMMARY:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose crossover bioavailability study on fenofibrate formulations comparing fenofibrate 160 mg tablets of Ranbaxy Laboratories with Tricor 160 mg tablets in healthy, adult, human subjects under fasting conditions.

DETAILED DESCRIPTION:
This was an open-label, randomized, single-dose, 2-way crossover, relative bioavailability study performed on 40 healthy adult male subjects.

As per protocol, enough healthy, adult, human subjects were to be enrolled in the study to allow the dosing of 40 subjects in the first period. 40 subjects were enrolled and a total of 37 subjects completed both the periods of study.

ELIGIBILITY:
Inclusion Criteria:

* Be in the age range of 18-45 years.
* Be neither overweight nor underweight for his/her height as per te Life insurance Corporation of india height/weight chart for non-medical cases.
* Have voluntarily given written informed consent to participate in this study.

Be of normal health as determined by medical history and physical examination of the subjects performed within 28 days prior to the commencement of the study.

If female and:

Of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence; or TS postmenopausal for at least 1 year; or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

History of allergy to fenofibrate and related fibric acid derivatives.

* History of gall stones/cholecystitis
* Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Presence of disease markers of H~-I and 2, Hepatitis B and C viruses and syphilis infection.

Female volunteers demonstrating a positive pregnancy screen.

Female volunteers who are currently breasffeeding.

* Presence of values which are clinically significantly different from normal reference ranges (as defined in Appendix 5) for haemoglobin, total white blood cells count, differential WBC count and platelet count.
* Positive for urinary screen testing of drugs of abuse (opiates and cannabinoids)
* Presence of values which are significantly different from normal reference ranges (as defined in Appendix 5) for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose, serum cholesterol and serum triglycerides.

Clinically abnormal chemical and microscopic examination of urine defined as presence .of RBC, WBC (>4/HPF), epithelial cells (>4/HPF), glucose (positive) and protein (positive).

Clinically abnormal ECG and Chest X-ray.

* History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma.
* History of any psychiatric illness which may impair the ability to provide written informed consent.
* Regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
* History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (! Unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or have difficulty in abstaining for the'duration of each study period.

Use of any enzyme modifying drugs within 30 days prior to Day 1 of this study.

Participation in any clinical trial within 6 weeks preceding Day ! of this study.

* Subjects who, through completion of this study, would have donated and/or lost more than 35;0 mL of blood in the past 3 months.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2002-11; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy Research Laboratories, Gurgaon, Haryana, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html